CLINICAL TRIAL: NCT02277678
Title: Comparison of Epidural Oxycodone and Epidural Morphine for Post Caesarean Section Analgesia: a Randomised Controlled Trial
Brief Title: Comparison of Epidural Oxycodone and Epidural Morphine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/321/D
Record Dates: First submitted 2014-10-26; First posted 2014-10-29 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Pruritus
Keywords: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone (Experimental): Epidural oxycodone 3mg single dose as opioid administration
  Interventions: Drug: Opioid administration oxycodone
- Morphine (Active Comparator): Epidural morphine 3mg single dose as opioid administration
  Interventions: Drug: Opioid administration morphine

INTERVENTIONS:
Drug: Opioid administration oxycodone — Epidural administration single dose through epidural catheter
  Other Names: Epidural Opioid
  Arms: Oxycodone
Drug: Opioid administration morphine
  Arms: Morphine

SUMMARY:
The primary objectives of this study are to compare the efficacy of pain relief between epidural oxycodone and epidural morphine for postoperative analgesia after elective caesarean section and to compare the incidence and severity of pruritus. Secondary objectives are to compare other side effects of epidural administered oxycodone and morphine (nausea and vomiting, sedation, respiratory depression) and to investigate the safety and efficacy of epidural oxycodone and epidural morphine after use for postoperative analgesia in caesarean sections.

DETAILED DESCRIPTION:
Undesirable side effects such as pruritus and nausea are common with epidural morphine and are thought to be due to mu-opioid receptor stimulation at the supra-spinal level. Recent studies of epidural oxycodone for abdominal and gynaecological surgery have shown that it is as effective as morphine with fewer side effects by this route. This has not been established in patients undergoing caesarean section. Oxycodone is a semi-synthetic opioid derivative that resembles morphine structurally and has similar lipid solubility. It has been reported that the analgesic action of oxycodone is more rapid in onset when compared with morphine and is mediated by kappa-opioid receptors in the spinal cord. The significance of our study would be to establish that epidural oxycodone reduces the side effects of pruritus of epidural morphine whilst still maintaining similar analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-2,
* aged between 21 to 50 years undergoing a term elective caesarean section and
* had consented for combined spinal-epidural (CSE) anaesthesia

Exclusion Criteria:

* concurrent opioid therapy,
* contraindications to CSE anaesthesia or any of the study medications,
* a history of pre-existing nausea and vomiting,
* failure to identify intrathecal space at time of anaesthesia,
* inadvertent dural puncture with the epidural needle and
* conversion of regional anaesthesia to general anaesthesia

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pruritus | 1 day
  Incidence of pruritus at 24 hours

SECONDARY OUTCOMES:
Pain | 1 day
  Pain score at 24 hours on using 0 to 10 scale
Nausea and Vomiting | 1 day
  Incidence of Nausea and Vomiting at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore, Singapore